CLINICAL TRIAL: NCT04278586
Title: Effect of Mindfulness on Opioid Use and Anxiety During Primary Care Buprenorphine Treatment (R33 Phase)
Acronym: Mindful-OBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHA-IRB-1114/06/19; R33AT010125 (NIH)
Record Dates: First submitted 2020-02-07; First posted 2020-02-20 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Opioid-use Disorder; Stress Related Disorder; Anxiety; Pain Interference
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two arms, live-online M-ROCC and live-online control, which are randomly assigned in a 1:1 ratio at the same time and are implemented in parallel.
Who Masked: Investigator
Masking Description: The principal investigator will be masked to arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live-Online Mindful Recovery OUD Care Continuum (Experimental): Live-Online Mindful Recovery OUD Care Continuum (M-ROCC) builds on other mindfulness interventions for addictive disorders, but is specifically designed for patients with OUD prescribed buprenorphine to be delivered in a live-online environment. It focuses on integration of mindfulness practice for living well through stress, anxiety, depression, pain and addiction recovery. The live-online M-ROCC curriculum has three primary components, including a low-dose mindfulness phase, an intensive mindfulness training phase and then a mindfulness maintenance check-in support group.
  Interventions: Behavioral: Live-Online M-ROCC
- Live-Online Control (Active Comparator): A time- and attention-matched live online control group. The manualized control intervention developed for the basic group-based opioid treatment group in primary care uses 16 core modules and 8 elective modules that are common to eclectic approach in treatment as usual addiction recovery groups (including engagement and group development activities with a mix of basic CBT skills, twelve-step facilitation, community reinforcement, and motivational interviewing). As an active group control, this method will help to isolate mindfulness as the putative mechanism of action by controlling for the therapeutic aspects of group without any reference to mindfulness.
  Interventions: Behavioral: Live-Online Control

INTERVENTIONS:
Behavioral: Live-Online M-ROCC — 1. LDM (Low-Dose Mindfulness): A 4-wk intro mindfulness program for OUD, 50-60 min/week including explicit training in use of mobile mindfulness apps, with rolling admission and ascending practice dose ladder.
  2. MTPC (Mindfulness Training for Primary Care): An eight-week intensive mindfulness group with ascending practice dose ladder and skill integration over 16 weeks with 60 minutes/wk.
  3. MCS (Mindfulness Maintenance Check-in Support): Ongoing weekly mindfulness group with check-in and reminders, leveraging mobile mindfulness apps and motivational counseling for graduates of LDM for 50-60 mins/wk.
  After completion of the LDM group, participation in various levels is fluid based on patient motivation, choice, and readiness.
  Arms: Live-Online Mindful Recovery OUD Care Continuum
Behavioral: Live-Online Control — A time- and attention-matched live online control group. The manualized control intervention developed for the basic group-based opioid treatment group in primary care uses 16 core modules and 8 elective modules that are common to eclectic approach in treatment as usual addiction recovery groups (including engagement and group development activities with a mix of basic CBT skills, twelve-step facilitation, community reinforcement, and motivational interviewing). As an active group control, this method will help to isolate mindfulness as the putative mechanism of action by controlling for the therapeutic aspects of group without any reference to mindfulness.
  Arms: Live-Online Control

SUMMARY:
This will be a randomized controlled trial (RCT) designed to compare live-online Mindful Recovery Opioid Care Continuum (M-ROCC) groups with a live-online control group on the primary outcome of number of biochemically confirmed opioid negative abstinent periods (defined by a negative oral fluid test [negative for opiate, oxycodone, fentanyl, methadone] AND no self-reported illicit opioid use) during the final six two-week periods of the study (study weeks 13-24).

DETAILED DESCRIPTION:
The investigators will conduct a RCT comparing Mindful Recovery Opioid Care Continuum (M-ROCC), a 24-week motivationally-responsive, trauma-sensitive, Group-Based Opioid Treatment (GBOT) program to a live-online control group, on the number of biochemically confirmed opioid negative abstinent periods (defined by a negative oral fluid test [negative for opiate, oxycodone, fentanyl, methadone] AND no self-reported illicit opioid use) during the final six two-week periods of the study (study weeks 13-24).

Clinical secondary outcomes include level of anxiety measured by the Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF), level of pain interference measured by the PROMIS Pain Interference Scale (PROMIS-PISF), and the number of positive oral fluid tests for BZD or cocaine during the final 12 weeks of the study. Other exploratory outcomes will be level of anxiety measured by the Beck anxiety inventory (BAI), 24-week intervention retention, as well as mechanisms of self-regulation assessed by self-report and behavioral measures (emotion regulation, decentering/metacognitive monitoring, interoception, experiential avoidance, self-critical rumination, and self-compassion) and their mediating effects on anxiety and opioid abstinence. Qualitative interviews will be conducted with a minimum of 12 and a maximum of 25 M-ROCC completers until thematic saturation to examine themes regarding live-online mindfulness delivery and to compare responses with our R21 qualitative outcomes from our in-person M-ROCC group model. Computerized Adaptive Testing for Mental Health (CAT-MH) will be used to assess changes in psychiatric co-morbidity. Finally, exploratory outcomes of stigma, mindfulness, perceived stress, pain catastrophizing, interpersonal conflict, and shared identity within group will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Participant lives in Massachusetts, Connecticut, Florida, Maine, New Hampshire, New York, Rhode Island, Texas, Vermont, California, Michigan, Illinois, North Carolina, Virginia, Arizona, and Alabama.
* Diagnosis of opioid use disorder prescribed a stable dose of buprenorphine (at least 4 weeks)
* Less than 90 days of abstinence (from non-prescribed opioids or benzodiazepines, cocaine, or alcohol) OR OUD with a co-morbid anxiety or stress disorder (as evaluated by Computerized Adaptive Testing for Mental Health [CAT-MH] or PROMIS-ASF > 55).
* Able to use an electronic device with a videocamera to attend study groups and complete questionnaires.
* Sufficient English fluency to understand procedures and questionnaires
* Ability to provide informed consent.

Exclusion Criteria:

* Active psychosis
* Bipolar I disorder history or severe level of mania on CAT-MH (>71)
* Acute suicidality or self-injurious behavior or severe level of suicidality on CAT-SS (>71)
* Cognitive inability as demonstrated by both the inability to complete an informed consent assessment AND complete the Montreal Cognitive Assessment Blind (MOCA BLIND) <24 on two different days
* Current participation in another experimental research study
* Previous participation in an 8-week intensive Mindfulness-Based Intervention in past 3 years or participation in the MINDFUL-OBOT pilot study
* Expected medical hospitalization in next 6 months
* Expected incarceration in next 6 months
* Substance use severity requiring likely inpatient treatment in opinion of principal investigator (e.g., severe alcohol withdrawal symptoms, severe benzodiazepine withdrawal symptoms, etc.).
* Inability to participate in group intervention without disrupting group in opinion of principal investigator or site PI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Cambridge Health Alliance, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosansky JA, Howard L, Goodman H, Okst K, Fatkin T, Fredericksen AK, Sokol R, Gardiner P, Parry G, Cook BL, Weiss RD, Schuman-Olivier ZD. Effects of live-online, group mindfulness training on opioid use and anxiety during buprenorphine treatment: A comparative effectiveness RCT. Contemp Clin Trials. 2024 Feb;137:107417. doi: 10.1016/j.cct.2023.107417. Epub 2023 Dec 20. PMID 38135210
- [Background] Fatkin T, Moore SK, Okst K, Creedon TB, Samawi F, Fredericksen AK, Roll D, Oxnard A, Le Cook B, Schuman-Olivier Z. Feasibility and acceptability of mindful recovery opioid use care continuum (M-ROCC): A concurrent mixed methods study. J Subst Abuse Treat. 2021 Nov;130:108415. doi: 10.1016/j.jsat.2021.108415. Epub 2021 Apr 15. PMID 34118705
- [Background] Schuman-Olivier Z, Fatkin T, Creedon TB, Samawi F, Moore SK, Okst K, Fredericksen AK, Oxnard AS, Roll D, Smith L, Cook BL, Weiss RD. Effects of a trauma-informed mindful recovery program on comorbid pain, anxiety, and substance use during primary care buprenorphine treatment: A proof-of-concept study. Am J Addict. 2023 May;32(3):244-253. doi: 10.1111/ajad.13364. Epub 2022 Dec 5. PMID 36470641
- [Background] Schuman-Olivier Z, Goodman H, Rosansky J, Fredericksen AK, Barria J, Parry G, Sokol R, Gardiner P, Le Cook B, Weiss RD. Mindfulness Training vs Recovery Support for Opioid Use, Craving, and Anxiety During Buprenorphine Treatment: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2454950. doi: 10.1001/jamanetworkopen.2024.54950. PMID 39836426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through Facebook, community partners (e.g., Lynn Community Health, Boston Medical Center, North Shore Community Health), online telemedicine providers (e.g., Bicycle Health, Boulder Care), and QR-code flyers linking an online referral form. Participants were recruited from 16 states including Massachusetts, Florida, Vermont, New Hampshire, Connecticut, New York, Maine, Texas, Rhode Island, California, North Carolina, Illinois, Michigan, Virginia, Alabama, and Arizona.
Pre-assignment Details: The PROMIS-ASF and CAT-MH was administered to participants after enrollment which may have caused participants to be excluded based on high mania or psychosis scores, low PTSD or anxiety scores, or no use in the past 90 days. Of 260 participants enrolled, 196 participants met the inclusion criteria and were randomized to begin the study.
Groups:
- Live-Online Mindful Recovery OUD Care Continuum: Live-Online Mindful Recovery OUD Care Continuum (M-ROCC) builds on other mindfulness interventions for addictive disorders, but is specifically designed for patients with OUD prescribed buprenorphine to be delivered in a live-online environment. It focuses on integration of mindfulness practice for living well through stress, anxiety, depression, pain and addiction recovery. The live-online M-ROCC curriculum has three primary components, including a low-dose mindfulness phase, an intensive mindfulness training phase and then a mindfulness maintenance check-in support group.
  Live-Online M-ROCC: 1. LDM (Low-Dose Mindfulness): A 4-wk intro mindfulness program for OUD, 50-60 min/week including explicit training in use of mobile mindfulness apps, with rolling admission and ascending practice dose ladder.
  2. MTPC (Mindfulness Training for Primary Care): An eight-week intensive mindfulness group with ascending practice dose ladder and skill integration over 16 weeks with 60 minutes/wk.
  3. MCS (Mindfulness Maintenance Check-in Support): Ongoing weekly mindfulness group with check-in and reminders, leveraging mobile mindfulness apps and motivational counseling for graduates of LDM for 50-60 mins/wk.
  After completion of the LDM group, participation in various levels is fluid based on patient motivation, choice, and readiness.
Period: Overall Study
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Started | 98 | 98
Completed | 48 | 68
Not Completed | 50 | 30
Not completed — Withdrawal by Subject | 13 | 6
Not completed — Lost to Follow-up | 37 | 24

BASELINE CHARACTERISTICS:
Population: This study used an intent-to-treat analysis model. Therefore, all participants that were randomized were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 95 | 192
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.4) | 40.9 (10.3) | 41.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 119
  Male | 38 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 88 | 91 | 179
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 90 | 90 | 180
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 4 | 7
Marital Status [Count of Participants; unit: Participants]
  Single | 43 | 44 | 87
  Married or Living as Married | 29 | 37 | 66
  Divorced | 18 | 14 | 32
  Widowed | 6 | 3 | 9
  Other | 2 | 0 | 2
Education (years) [Mean (Standard Deviation); unit: years] | 13.1 (2.2) | 13.5 (2.6) | 13.3 (2.4)
Sexual Identity [Count of Participants; unit: Participants]
  Straight or Heterosexual | 81 | 78 | 159
  Lesbian, Gay, or Homosexual | 3 | 6 | 9
  Bisexual | 9 | 10 | 19
  Other | 5 | 4 | 9
Annual Income [Count of Participants; unit: Participants]
  <$20,000 | 37 | 46 | 83
  $20,000-$80,000 | 53 | 38 | 91
  >$80,000 | 7 | 14 | 21
  Unreported | 1 | 0 | 1
Buprenorphine Dose [Mean (Standard Deviation); unit: milligrams] | 13.3 (6.3) | 15.7 (6.9) | 14.5 (6.7)
Opioid Craving Scale [Mean (Standard Deviation); unit: units on a scale] — Scale Range 0-30, higher rating meant greater craving and vice versa.
  units on a scale | 3.4 (2.5) | 3.0 (2.5) | 3.2 (2.5)
Unemployment Status [Count of Participants; unit: Participants] | 18 | 17 | 35
Participants with 4+ Adverse Childhood Events (ACES) [Count of Participants; unit: Participants] | 65 | 65 | 130
Patient-Reported · Outcomes Measurement Information System (PROMIS)-Anxiety T-Score [Mean (Standard Deviation); unit: T-score] — The mean of the T score is 50 with a standard deviation of 10. Higher scores represent greater anxiety and vice versa. This study determined a T score of 55 to indicate elevated anxiety.
  T-score | 64.5 (6.2) | 65.9 (6.8) | 65.2 (6.5)
Patient-Reported · Outcomes Measurement Information System (PROMIS)-Pain Interference T-Score [Mean (Standard Deviation); unit: T-score] — The mean of the T score is 50 with a standard deviation of 10. Higher scores represent greater pain interference and vice versa. This study determined a T score of 55 to indicate elevated pain interference.
  T-score | 60.9 (9.0) | 59.1 (10.1) | 60.0 (9.6)
Lifetime heroin use [Count of Participants; unit: Participants] | 56 | 59 | 115
Lifetime cocaine or crack use [Count of Participants; unit: Participants] | 78 | 67 | 145
Used fentanyl in 90 days before screening [Count of Participants; unit: Participants] | 8 | 3 | 11
Past mindfulness experience [Count of Participants; unit: Participants] | 17 | 21 | 38
Region of the US [Count of Participants; unit: Participants]
  Northeast | 24 | 27 | 51
  South | 48 | 47 | 95
  Midwest | 14 | 10 | 24
  West | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Biochemically-confirmed Opioid Abstinent 2-week Time Periods
Description: Biochemically-confirmed opioid abstinence, which is defined as the number of two-week periods with a negative oral fluid screen AND no opioid use reported in weekly self report self-report during the final 12 weeks (weeks 13-24) of the study (6 is the highest possible number of negative oral fluid toxicology screen time periods). Participants will be randomly selected to undergo a live-online supervised oral fluid screen at a rate of once every 2 weeks.
Time Frame: Weeks 13-24
Population: Using an intent-to-treat, mixed-effects GEE analysis with the covariates baseline buprenorphine dose, cocaine use, and annual income.
Measure: Mean (95% Confidence Interval); unit: percentage of 2-week time periods
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
percentage of 2-week time periods | 13.4 [6.2 to 20.5] | 12.7 [7.5 to 18.0]

2. Secondary Outcome: Number of Positive Oral-fluid Toxicology Tests for Cocaine.
Description: Biochemically-confirmed cocaine use, which is defined as the number of two-week periods with a positive oral-fluid screen. Oral-fluid toxicology screens will be conducted during the final 12 weeks (weeks 13-24) of the study (6 is the highest possible number of negative oral fluid toxicology screen time periods). Participants will be randomly selected to undergo a live-online supervised oral fluid screen at a rate of once every 2 weeks.
Time Frame: Weeks 13-24
Population: We used an intent-to-treat approach, mixed-effects GEE analysis with the covariates baseline buprenorphine dose, cocaine use, and annual income.
Measure: Mean (95% Confidence Interval); unit: percentage of 2-week time periods
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
percentage of 2-week time periods | 8.4 [0 to 16.6] | 1.5 [0 to 4.0]

3. Secondary Outcome: Number of Positive Oral-fluid Toxicology Tests for Benzodiazepines.
Description: Biochemically-confirmed benzodiazepine use, which is defined as the number of two-week periods with a positive oral-fluid screen. Oral-fluid toxicology screens will be conducted during the final 12 weeks (weeks 13-24) of the study (6 is the highest possible number of negative oral fluid toxicology screen time periods). Participants will be randomly selected to undergo a live-online supervised oral fluid screen at a rate of once every 2 weeks.
Time Frame: Weeks 13-24
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of 2-week time periods
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
percentage of 2-week time periods | 22.1 [12.7 to 31.5] | 20.2 [12.7 to 27.7]

4. Secondary Outcome: Patient Report Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF)
Description: The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale from 7-35 used to assess patient-reported health status for anxiety. Subjects are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always). Higher ratings indicate greater anxiety symptoms while lower ratings indicate less anxiety symptoms. This will be assessed among participants with an anxiety disorder (defined as PROMIS >55 at baseline) as well at weeks 8, 16, and 24.
Time Frame: 24 Weeks
Population: Difference-in-differences, intent-to-treat, repeated measures analysis using linear mixed effects models with a study week by group interaction term to estimate the relative changes from baseline to week 24. We included only those participants with PROMIS-ASF T-scores above 55 at baseline.
Measure: Mean (95% Confidence Interval); unit: differences in scores on a scale
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
differences in scores on a scale | -9.0 [-11.7 to -6.3] | -10.0 [-12.0 to -8.0]

5. Secondary Outcome: Pain Interference PROMIS (PROMIS-PISF)
Description: The PROMIS Pain Interference instruments measure the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. The Pain Interference short form is universal rather than disease-specific. It assesses pain interference over the past seven days. Each question has five response options ranging in value from one to five with a total scale range of 7-35. Higher ratings indicate greater pain interference and lower ratings indicate lesser pain interference. This assessment was done at baseline and weeks 8, 16, and 24.
Time Frame: 24 Weeks
Population: Difference-in-differences, intent-to-treat, repeated measures analysis using linear mixed effects models with a study week by group interaction term to estimate the relative changes from baseline to week 24.
Measure: Mean (95% Confidence Interval); unit: differences in scores on a scale
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
differences in scores on a scale | -4.1 [-7.3 to -0.9] | -4.4 [-6.8 to -2]

6. Other Pre Specified Outcome: Substance Craving Scale (SUBCS)
Description: The Substance Craving Scale (SUBCS) is a 6-item scale with a range of 0-60. It includes the 3-item validated Opioid Craving Scale (OCS) as the primary measure with a 0-30 scale based on opioids. The SUBCS adds another 3 items based on other non-opioids substances. The OCS assesses participant craving for Opioids (including fentanyl, heroin, methadone, oxycodone or other opioids) and the (SUBCS) includes the OCS plus other substance use (including illicit drugs [e.g., cocaine, methamphetamine, etc.], using unprescribed pills or prescribed medications in ways or at doses for which they were not prescribed [e.g., Klonopin, etc.], or drinking alcohol). This study uses the 3-items specifically from the Opioid Craving Scale (OCS) as our outcome measure for this study with a range of 0-30 and includes SUBCS as exploratory. Higher ratings on OCS indicate greater opioid craving and lower ratings indicate less opioid craving.
Time Frame: 24 Weeks
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
Number analyzed (Participants) | 98 | 98
score on a scale | -2.3 [-2.9 to -1.7] | -1.3 [-1.9 to -0.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 24 weeks that participants were in the study.
Description: The definitions do not differ. Staff monitored adverse events (AEs) at each study visit and via a REDCap survey at weeks 8, 16, and 24, rated by severity, relatedness, expectedness, with regular DSMB review. All-Cause Mortality was not monitored/assessed.
Arm/Group | Live-Online Mindful Recovery OUD Care Continuum | Live-Online Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 7/98 | 2/98
Other Adverse Events (participants affected / at risk) | 29/98 | 21/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Live-Online Mindful Recovery OUD Care Continuum (N=98) | Live-Online Control (N=98)
Infection (Infections and infestations) | 3 | 0 — Pt hospitalized for infection in chin. Not related to study. Pt hospitalized for infection in blood. Needed IV antibiotics. Not related to study. Participant was hospitalized for poison ivy infection. Not related to study.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Lung issues related to pneumonia. Not related to the study.
Heart and Lung Problems (Cardiac disorders) | 0 | 1 — Heart and lung problems. Patient was hospitalized for a couple of days. Not related to the study.
Overdose (Psychiatric disorders) | 1 | 0 — Vomited and swallowed vomit while sleeping due to overconsumption of CBD gummies. Not study related. Was hospitalized for a few days.
Covid-19 (Immune system disorders) | 1 | 0 — Participant was hospitalized due to Covid-19 symptoms. Not study related.
Surgery (Surgical and medical procedures) | 0 | 1 — Participant had to have emergency surgery to remove their gallbladder after feeling pain. Not study related.
Miscarriage (Reproductive system and breast disorders) | 1 | 0 — Participant had a miscarriage that required surgery. Not related to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Live-Online Mindful Recovery OUD Care Continuum (N=98) | Live-Online Control (N=98)
Sickness (Immune system disorders) | 2 | 3 — Participants experienced cold symptoms. Not study related.
Developed a new condition (General disorders) | 5 | 1 — Participants developed new conditions. Not study related
Worsening Psychiatric Symptoms/Stress (Psychiatric disorders) | 7 | 5 — Participants experienced an increase in anxiety, depression, and/or stress. Not study related
Pain (General disorders) | 4 | 5 — Participants experienced increases in pain symptoms. Not study related.
Stomach Issues (Gastrointestinal disorders) | 2 | 1 — Participants experienced stomach pain or gastrointestinal issues. Not study related
Injury (Injury, poisoning and procedural complications) | 3 | 2 — Participants experienced injuries. Not study related.
Headaches (Nervous system disorders) | 2 | 0 — Participants experienced headache symptoms. Not study related.
Cardiac Issues (Cardiac disorders) | 1 | 0 — Participant experienced heart issues. Not study related.
Kidney stones (Renal and urinary disorders) | 1 | 1 — Participants experienced kidney stones. Not study related.
Pain (General disorders) | 1 | 0 — Participant experienced pain during a mindfulness practice. This was related to the study.
Relapse (Psychiatric disorders) | 1 | 0 — Participant experienced a relapse in their drinking. Not study related.
Pregnancy (Reproductive system and breast disorders) | 0 | 3 — Participants experienced symptoms related to their pregnancies. Not study related.

LIMITATIONS AND CAVEATS:
1. The study had higher attrition levels for M-ROCC than a prior study between during weeks 8-16 after a warning about the increased intensity and trauma-informed choice to remain in group.
2. This study had an evidence-based active comparator and lacked a control condition with no behavioral treatment.
3. The predominantly White sample reflects national trends in buprenorphine treatment engagement and existing disparities in equitable treatment access, but limits study generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT04278586/Prot_SAP_006.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT04278586/ICF_007.pdf